CLINICAL TRIAL: NCT01641445
Title: Effects of Topiramate on Adolescent Alcohol Use: Efficacy and Mechanisms
Acronym: IMPACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Robert Miranda, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AA007850-21 (NIH)
Record Dates: First submitted 2012-07-11; First posted 2012-07-16 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Active Comparator): Topiramate (200 mg) taken orally daily
  Interventions: Drug: Topiramate
- Sugar pill (Placebo Comparator): Placebo ("sugar pill") taken orally daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate (200 mg daily)
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Matching placebo capusules ("sugar pills"
  Other Names: "Sugar Pill"
  Arms: Sugar pill

SUMMARY:
This study will help to determine whether the medication, topiramate, reduces alcohol use among adolescents with alcohol dependence. It will also help answer the question, "How does topiramate reduce drinking in teenagers?" Understanding how topiramate may reduce drinking in adolescents would allow for a more targeted pharmacotherapeutic approach to treatment and help to identify additional medications that may hold promise for improving treatment outcomes for youth.

DETAILED DESCRIPTION:
Adolescent alcohol use is associated with myriad adverse legal, health, and educational consequences and contributes to the leading causes of mortality among youth. Yet despite the magnitude of this public health problem, treatment initiatives for youth remain inadequate. Given these data, the National Institute on Alcohol Abuse and Alcoholism identified the critical need for medications development research for youth with the goal of identifying promising agents for which large-scale clinical trials are justified. The long-term goal of this research program is to improve pharmacotherapy for alcoholism. The major objective of this project is to address the urgent need for empirical data on medications that may benefit youth. For the past 10 years our research program has successfully paired human laboratory paradigms with ecological momentary assessment (EMA), whereby research participants use handheld electronic diaries to monitor their drinking, craving, and sensitivity to alcohol in real time in their natural environment. Using this approach, we identified mechanisms by which medications act and patient characteristics that moderate these effects. The proposed study will test if and how topiramate (TPM), an anticonvulsant shown to be efficacious for treating adults, reduces drinking in youth. To this end, we will randomize adolescent problem drinkers to TPM or placebo for 8 weeks, in combination with biweekly motivational enhancement therapy sessions, using a two-group, double-blind design. While at the target dose (200 mg/day) youth will complete EMA in their natural environment. In addition, youth will complete alcohol cue reactivity assessments in the laboratory to test the effects of TPM on cue-elicited craving and physiological reactivity in a controlled environment. Youth will complete 6- and 12-month follow-up assessments to determine whether any benefits are sustained. This study will provide much needed data on the tolerability and efficacy of TPM with adolescents, while adding important new information about the biobehavioral mechanisms of TPM action in youth.

ELIGIBILITY:
Inclusion Criteria:

* 14-24 years old (inclusive)
* Non-treatment seeking for alcohol abuse or dependence
* Interest in reducing alcohol use
* Self-reported alcohol use at least 2 days/week during prior 28 days
* Able to read simple English

Exclusion Criteria:

* Alcohol or substance abuse treatment in the past 30 days
* Clinically significant medical abnormalities
* History of renal impairment, renal stones, or unstable hypertension
* History of progressive neurodegenerative disorders or clinical significant neurological disorders
* Body mass index lower than 18
* Pregnant, nursing, or refusal to use reliable birth control, if female
* Non-stabilized psychotropic medication and/or taking medication that is contraindicated for use with topiramate
* Medications that may effect alcohol use or a carbonic anhydrase inhibitor
* Suicidal or psychotic
* Current coexisting substance use disorders other than alcohol, caffeine, cannabis, or nicotine use disorders
* Clinically significant alcohol withdrawal symptoms
* Impaired cognitive functioning
* Living with an active study participant
* Compelled to treatment by the juvenile justice system

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miranda, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Sugar Pill
Started | 41 | 41
Completed | 31 | 36
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Sugar Pill | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.88 (2.08) | 20.49 (2.05) | 20.68 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 21 | 21 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Percent drinking days at the target medication dose
Time Frame: Study Weeks 5-8
Measure: Mean (Standard Deviation); unit: Percent of days
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 41 | 41
Percent of days | 29.59 (19.55) | 27.08 (21.47)

2. Primary Outcome: Heavy Drinking Days
Description: Percent heavy drinking days at the target medication dose. Heavy drinking is defined as 4 or more standard alcoholic drinks per day for females and 5 or more standard drinks per day for males.
Time Frame: Study Weeks 5-8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 41 | 41
percentage of days | 9.34 (10.99) | 6.78 (11.44)

3. Secondary Outcome: Alcohol Use
Description: Percent drinking days at the 6-month follow-up assessment
Time Frame: 6-month follow-up assessment
Measure: Mean (Standard Deviation); unit: Percent of days
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 24 | 31
Percent of days | 23.56 (17.11) | 21.75 (21.50)

4. Secondary Outcome: Alcohol Use
Description: Percent drinking days at the 12-month follow-up assessment
Time Frame: 12-month follow-up assessment
Measure: Mean (Standard Deviation); unit: Percent of days
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 22 | 27
Percent of days | 25.55 (22.03) | 21.93 (21.73)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 8-week active medication (or placebo pill) period.
Description: The definitions of adverse event and serious advserse event are the same as those used by clinicaltrials.gov.
Arm/Group | Topiramate | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 37/41 | 35/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=41) | Sugar Pill (N=41)
Slow Thinking or Reactions (General disorders) | 12 | 3
Nervousness (Psychiatric disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 14 | 4
Difficulty with Memory (Psychiatric disorders) | 12 | 4
Word Finding Difficulties (Psychiatric disorders) | 13 | 3
Fatigue (General disorders) | 12 | 8
Difficulty with Concentration or Attention (Psychiatric disorders) | 13 | 3
Depression (Psychiatric disorders) | 4 | 1
Confusion (Psychiatric disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 10 | 10
Weight Loss (General disorders) | 13 | 11
Decrease in Appetite (General disorders) | 13 | 6
Paresthesias (General disorders) | 22 | 2
Eye Problems (Eye disorders) | 6 | 2
Changes in Vision (Eye disorders) | 6 | 2
Runny Nose, Sinus Problems, Sneezing (General disorders) | 14 | 17
Injuries (General disorders) | 5 | 7
Headache (General disorders) | 12 | 13
Sore Throat (General disorders) | 10 | 8
Diarrhea (Gastrointestinal disorders) | 3 | 0
Elevated Heart Rate (General disorders) | 4 | 0
Stomach Discomfort (Cramps/Bloated) (General disorders) | 4 | 0
Fever (General disorders) | 3 | 0
Cough (General disorders) | 8 | 9
Dizziness (General disorders) | 12 | 1
Difficulty with Coordination or Balance (General disorders) | 6 | 1
Drowsiness or Sleepiness (General disorders) | 16 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT01641445/ICF_000.pdf